CLINICAL TRIAL: NCT05874427
Title: Comparison of Patient Understanding and Anxiety Between the New Imaging Consent Form and the Existing Narrative Consent Form When Explaining the Procedure Pilot Study
Brief Title: Comparison Between the Imaging Consent Form and the Existing Narrative Consent Form
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Pyung-Bok Lee, Principal Investigator, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: B-2206-761-303
Record Dates: First submitted 2023-05-10; First posted 2023-05-24 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2024-04

CONDITIONS: Lumbar Radiculopathy
Keywords: lumbar radiculopathy; Multimedia informed consent
MeSH Terms: conditions — Radiculopathy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multimedia informed consent (Experimental): Multimedia informed consent with videos to explain transforaminal epidural steroid injection
  Interventions: Procedure: Multimedia informed consent
- Standard informed consent (Active Comparator): A standard consent form to describe the procedure previously used.
  Interventions: Procedure: Standard informed consent

INTERVENTIONS:
Procedure: Multimedia informed consent — A standard consent form on paper to explain the procedure, with an additional video to explain the procedure and risks.
  Arms: Multimedia informed consent
Procedure: Standard informed consent — A standard consent form, written on paper, used to explain a procedure to a patient face-to-face by a physician.
  Arms: Standard informed consent

SUMMARY:
This is a single-center, randomized, double-blind clinical study to compare patient comprehension and anxiety by comparing a traditional paper consent form to a multimedia consent form for patients undergoing transforaminal epidural steroid injection.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Patients undergoing lumbar transforaminal block for the first time
* Patients who are able to understand the contents of the video consent form and written consent form.

Exclusion Criteria:

* Patients who have difficulty understanding or answering consent forms
* Patients who have previously experienced a transforaminal steroid injection

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2023-05-22 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2023-10-01 (Actual)

PRIMARY OUTCOMES:
Patient comprehension assessed by Patient comprehension questionnaire | immediately before the procedure
  A questionnaire to assess the understanding of the procedure in patients undergoing transforaminal epidural steroid injections, created by three pain medicine specialists. The test consists of 10 questions, all of which are answered with a yes/no response to provide a score from 0 to 10.

SECONDARY OUTCOMES:
Anxiety assessed by Spielberger State-Trait Anxiety Inventory (STAI) short form | immediately before the procedure
  used to measure the state and trait components of anxiety The test consists of six questions, each of which is scored on a scale from not at all (1) to very much so (4), depending on the patient's response. Scores range from 6 to 24, with lower scores indicating higher anxiety state.
Assess patient satisfaction by Patient satisfaction ratings on a Likert scale | immediately after the procedure
  Patient satisfaction ratings on a Likert scale The test consists of five questions, each of which is answered on a scale from not at all (0) to very much so (4), depending on the patient's response. Scores range from 0 to 20, with higher scores indicating better understanding.

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul national university Bundang hospital, Seongnam, Kyoungki-do, South Korea